CLINICAL TRIAL: NCT05716503
Title: Comparison Between Negative Pressure Wound Therapy and Conventional Wound Dressings Before and After Split-Thickness Skin Grafting in Diabetic Foot Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hady Khaled Elhossiny, Resident of plastic and reconstructive surgery, Sohag University hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Soh-Med-23-01-08
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Negative-Pressure Wound Therapy; Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Patients will randomly be divided into two groups - study group and control group. Study group (A): Will Receive negative pressure wound therapy dressings before skin grafting to prepare the wound bed and after skin grafting.
  Control group (B): Will Receive once daily dressing with antibiotic ointment and gauze before and after skin grafting.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (A) (Experimental): Study group (A): Will Receive negative pressure wound therapy dressings before skin grafting to prepare the wound bed and after skin grafting.
  Interventions: Device: Negative Pressure Wound Therapy (NPWT)
- Control group (B) (Experimental): Control group (B): Will Receive once daily dressing with antibiotic ointment and gauze before and after skin grafting.
  Interventions: Other: Ordinary dressings with antibiotic ointment and gauze

INTERVENTIONS:
Device: Negative Pressure Wound Therapy (NPWT) — Patients Will Receive negative pressure wound therapy dressings before skin grafting to prepare the wound bed and after skin grafting.
  Arms: Study group (A)
Other: Ordinary dressings with antibiotic ointment and gauze — Patients will Receive once daily dressing with antibiotic ointment and gauze before and after skin grafting.
  Arms: Control group (B)

SUMMARY:
The aim of this thesis is to compare the efficacy of Vacuum assisted closure device versus conventional dressing before and after split thickness skin grafting in diabetic foot wounds.

DETAILED DESCRIPTION:
Negative pressure wound therapy is a new noninvasive technique for treating open wounds. It works by removing fluid from the wound bed, reducing edema, and encouraging the growth and perfusion of new granulation tissue.

Vacuum-Assisted Closure device (VAC) helps to remove fluid from open wounds through a sealed dressing and tubing which is connected to a collection container. Vacuum-assisted closure (VAC) can provide stable and persistent negative pressure, and there are several modes to choose from.

VAC has played an important role in helping to close wounds, controlling infection, promoting angiogenesis, increasing blood flow, and promoting granulation tissue growth in wounds. It is now widely applied in all kinds of acute, chronic, and special wounds with good therapeutic results. However, there is a need to pay attention to contraindications and complications of VAC when it is used, avoiding secondary damage due to improper treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age group 20-75 years.
* Patients with diabetic foot wounds who are scheduled for skin grafting.

Exclusion Criteria:

* Age <20 years or > 75 years.
* An obvious septicemia.
* Foot osteomyelitis.
* Ulcer resulting from venous insufficiency.
* Features of malignant ulcer.
* Patients being treated with corticosteroids, immunosuppressive drugs.
* Any other serious pre-existing cardiovascular, pulmonary or immunological disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Period of hospitalization. | 2 weeks
  Number of days of patient hospitalization before and after grafting
Time of complete healing | 1 month
  Number of days needed for each patient for complete healing after operation
Functional outcome | 5 months
  Number of patients with full range of mobility at site of graft Vs number of patients with limited mobility
Patient satisfaction of aesthetic outcome | 5 months
  Number of patients satisfied with the aesthetic result of the operation on a scale of 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sinha K, Chauhan VD, Maheshwari R, Chauhan N, Rajan M, Agrawal A. Vacuum Assisted Closure Therapy versus Standard Wound Therapy for Open Musculoskeletal Injuries. Adv Orthop. 2013;2013:245940. doi: 10.1155/2013/245940. Epub 2013 Jun 26. PMID 23878741
- [Background] Lone AM, Zaroo MI, Laway BA, Pala NA, Bashir SA, Rasool A. Vacuum-assisted closure versus conventional dressings in the management of diabetic foot ulcers: a prospective case-control study. Diabet Foot Ankle. 2014 Apr 8;5. doi: 10.3402/dfa.v5.23345. eCollection 2014. PMID 24765245
- [Background] Ali Z, Anjum A, Khurshid L, Ahad H, Maajid S, Dhar SA. Evaluation of low-cost custom made VAC therapy compared with conventional wound dressings in the treatment of non-healing lower limb ulcers in lower socio-economic group patients of Kashmir valley. J Orthop Surg Res. 2015 Dec 10;10:183. doi: 10.1186/s13018-015-0314-5. PMID 26654318
- [Background] Ravari H, Modaghegh MH, Kazemzadeh GH, Johari HG, Vatanchi AM, Sangaki A, Shahrodi MV. Comparision of vacuum-asisted closure and moist wound dressing in the treatment of diabetic foot ulcers. J Cutan Aesthet Surg. 2013 Jan;6(1):17-20. doi: 10.4103/0974-2077.110091. PMID 23723599